CLINICAL TRIAL: NCT07296835
Title: Surgical Outcomes and Costs in Using the Shenzhen HugeMed 6.3 French Flexible Ureteroscope
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00161756
Record Dates: First submitted 2025-12-04; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Kidney Stones
Keywords: hugemed, coast saving, ureteroscopy
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Intervention Model Description: This study employs a hybrid design: a prospective single-arm cohort of patients undergoing RIRS, with outcomes measured at predefined intervals. To provide comparative context, a retrospective control cohort will be identified from KUMC's electronic medical records of patients who also underwent RIRS by SOC with traditional f-URS scope, matched 2:1 based on key baseline characteristics (e.g., age, sex, stone size, etc.). This will allow for retrospective comparison of outcomes between the intervention group and standard management
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- hugemed ureteroscopy (Active Comparator): Patients scheduled to undergo URS retrograde intrarenal surgery per standard of care will be recruited from urology clinics or OR schedules using using the 6.3 Fr f-URS . Patients may be approached and consented in clinic or pre-op.
  All procedures, devices, and ancillary equipment are standard of care. There is no additional cost to the patient, only the typical standard of care costs. Participants will not be compensated for participation in the study.
  Interventions: Device: Ureteroscopy using the 6.3 Fr f-URS hugemed; Device: Hugemed 6.3 Fr f-URS

INTERVENTIONS:
Device: Ureteroscopy using the 6.3 Fr f-URS hugemed — All patients will be counseled on standard treatment options. Treatment options and subsequent care will not deviate from routine care. If they do not enroll in the study, the HU30M may still be used during routine surgery and care. The only intervention specific to the research will involve the use of patient information in describing the results. Participants will undergo RIRS in standard fashion, without deviation from the standard of care. Patients will be brought to the operating room, positioned, and placed under general anesthesia. RIRS will be performed using HU30M 6.3 Fr f-URS. Laser platform (ex: HoYAG or TFL) as well as laser settings will be at the treating investigator's discretion and may be changed during the procedure at their discretion as well, all per standard of care. The initial laser settings and changes that occurred to the settings after the first minute of the case will be recorded.
Device: Hugemed 6.3 Fr f-URS — Retrograde intrarenal surgery will be performed using HU30M 6.3 Fr f-URS.

SUMMARY:
Comprehensive comparative investigations between HugeMed HU30M 6.3 Fr f-URS and traditional approach f-URS devices in RIRS are lacking in an American population. The investigators aim to compare the outcomes of using the 6.3 Fr f-URS versus traditional approach (other f-URS present in our institution) to treat patients with stone burden ≤ 2.5 cm. The findings of this study will expand on the potential advantages and drawbacks of HU30M in enhancing surgical outcomes and patient safety in RIRS procedures. We hypothesize that the use of the HU30M will result in increased cost savings while providing similar stone free rates when compared to traditionally used f-URS devices.

ELIGIBILITY:
Inclusion Criteria:

* Males or females ³ 18 years of age
* Patients with ureteral or kidney stones undergoing primary flexible ureteroscopy for retrograde intrarenal surgery
* Total stone burden ≤ 2.5 cm

Exclusion Criteria:

* Undergoing bilateral stone treatment during the same procedure
* Patients with known genitourinary anatomical abnormalities that would complicate the procedure as determined by the treating investigator
* Uncorrected coagulopathy
* Patients with urinary diversions
* Chronic external urinary catheters
* Women who are pregnant
* Immunosuppressed patients
* Non-elective procedures
* Participants must not be involved in any other clinical research studies during the duration of this trial. Exceptions may be made if the investigator determines, on a case-by-case basis, that participation in another study will not adversely affect the outcomes or integrity of this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
To evaluate and compare outcomes and costs associated with hugeMed 6.3 Fr flexible URS versus traditional approach in RIRS | 36 months
  Stone free rate, defined as the absence of residual stone fragments > 2 mm, as determined by noncontrast CT scan performed

CONTACTS AND LOCATIONS:
Overall Officials: Wilson R. Molina, md, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University Of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No
data will be used to compare different outcomes from ureteroscopy surgeries